CLINICAL TRIAL: NCT05625802
Title: Erector Spinae Plane Block for Uncomplicated Renal Colic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Christopher Fung, Assistant Professor in Emergency Medicine - Adult, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00219913
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Renal Colic; Kidney Stone
Keywords: erector spinae plane block; Emergency Department; ropivacaine
MeSH Terms: conditions — Renal Colic; Kidney Calculi; Emergencies | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Single site two-stage open label phase 2 clinical trial with one treatment arm and one external control arm
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erector Spinae Plane Block (ESPB) (Experimental): Intervention inhibits neurotransmission at the dorsal and ventral rami of the thoracic spinal nerves, providing anesthesia to multiple dermatomal levels
  Interventions: Procedure: Erector Spinae Plane Block (ESPB); Drug: Ropivacaine
- External control (No Intervention): External control patients will be selected from a population of patients meeting the following criteria: 1) adult ED patient with the diagnosis of uncomplicated kidney stones; 2) received at least one dose of parenteral medication while in the ED; 3) presentation to the ED between 7/1/2021 and the study start date. From this population, propensity score matched control patients will be selected at a ratio of 3 controls to 1 ESPB patient. External control population patients are not active patients in this study and analysis of their data will be secondary use of data collected during routine care.

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (ESPB) — Up to 30 Cubic Centimeter (cc) of 0.5% ropivacaine administered by local injection into the erector spinae plane under ultrasound guidance
  Arms: Erector Spinae Plane Block (ESPB)
Drug: Ropivacaine — 0.5% ropivacaine
  Arms: Erector Spinae Plane Block (ESPB)

SUMMARY:
This research study is to determine how well the Erector Spinae Plane Block (ESPB) works for kidney stone pain and any possible side effects.

DETAILED DESCRIPTION:
When this trial was initially started, the intent was to compare the Erector Spinae Plane Block (ESPB) arm to data from electronic health records (EHR) of patients who had not received the ESPB. The EHR data was never obtained, so no comparison was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Imaging confirmation of urolithiasis on the index encounter or prior encounter within 7 days
* Patient received one dose of parenteral pain medication in the emergency department (ED)

Exclusion Criteria:

* Pregnancy or breastfeeding
* Prisoner or incarcerated individual
* Therapeutic anticoagulation or coagulopathy.
* Active treatment for urinary tract infection (either acute infection or chronic therapy)
* Prior spinal surgery in the thoracic region
* Allergy to local anesthetic or prior local anesthetic
* Soft tissue infection overlying the injection site
* Positive for coronavirus
* Inability to communicate verbally or read/write in English
* Currently taking strong CYP1A2 inhibitor (fluvoxamine, amiodarone, fluoroquinolones, etc.)
* Glucose-6-phosphate dehydrogenase deficiency (G6PD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Fung, Study Chair — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: When this trial was initially started, the intent was to compare the Erector Spinae Plane Block (ESPB) arm to data from electronic health records (EHR) of patients who had not received the ESPB. The EHR data was never obtained, so no comparison was conducted.
Groups:
- External control: Control patient data (external controls that did not receive ESPB), routinely collected health information, collected as secondary data.
Period: Overall Study
Arm/Group | Erector Spinae Plane Block (ESPB) | External control
Started | 5 | 0
Completed | 4 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erector Spinae Plane Block (ESPB)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
First paraenteral pain medicine [Count of Participants; unit: Participants] — Initial paraenteral pain medicine taken by participants.
  Participants
    Ketorolac | 4
    Morphine | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Received a Second Parenteral Pain Medication in the Emergency Department (ED)
Description: Results reflect the number of participants who received a second parenteral pain medication after receiving one already. Data for this outcome was collected via electronic health record query.
Time Frame: By ED discharge, approximately 12 hours or less
Measure: Count of Participants; unit: Participants
Arm/Group | Erector Spinae Plane Block (ESPB)
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Change in Pain
Description: Pain ranked on a visual analog scale of 1-10, where 10 indicated the most pain and 1 indicated no pain. Change was defined as the last pain score minus first pain score.
Time Frame: Baseline, 5 minutes, and 60 minutes following procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erector Spinae Plane Block (ESPB)
Number analyzed (Participants) | 5
score on a scale
  Baseline | 3.2 (3.1)
  5 minutes following | 1.8 (1.8)
  60 minutes following procedure | 1.8 (1.8)

3. Secondary Outcome: Rate of Admission to Hospital for Kidney Stones
Description: Results reflect participants who were admitted to the hospital for kidney stones at or prior to day 7 and at or prior to day 30 following administration of the intervention. Data for this outcome was collected via electronic health record query.
Time Frame: Up to 30 days
Population: Data was only collected for participants who were still in the trial by day 7 and day 30. 1 participant was lost to follow up before day 30.
Measure: Count of Participants; unit: Participants
Arm/Group | Erector Spinae Plane Block (ESPB)
Number analyzed (Participants) | 5
Participants
  7 days | 2
  30 days: number analyzed (Participants) | 4
  30 days | 1

4. Secondary Outcome: Rate of 24-hour and 72-hour Return to the Emergency Department (ED)
Description: Results reflect participants who returned to the ED for kidney stone-related issues at 24 hours and 72 hours following administration of the intervention. Data for this outcome was collected via electronic health record query.
Time Frame: Up to 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Erector Spinae Plane Block (ESPB)
Number analyzed (Participants) | 5
Participants
  24 hours | 0
  72 hours | 0

5. Secondary Outcome: Emergency Department Length of Stay
Description: Average length of stay in the emergency department per participant.
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Erector Spinae Plane Block (ESPB)
Number analyzed (Participants) | 5
minutes | 418 (183)

6. Secondary Outcome: Safety Outcomes and Complications
Description: Results reflect the number of participants who were still in the trial by day 30 and had experienced any of the pre-defined safety events.
Time Frame: Up to 30 days
Population: 1 participant was lost to follow up prior to Day 30.
Measure: Count of Participants; unit: Participants
Arm/Group | Erector Spinae Plane Block (ESPB)
Number analyzed (Participants) | 4
Participants
  Admission to hospital due to nerve block complication | 0
  Injury to a blood vessel that is permanent | 0
  Injury to a nerve that is permanent | 0
  Injury to blood vessel that required surgery | 0
  Injury to lung that required surgery | 0
  Infection of the skin, muscle of soft tissue of back | 0
  Allergic reaction to medicine used for nerve block | 0
  Other reaction to medicine used for nerve block | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days
Description: When this trial was initially started, the intent was to compare the Erector Spinae Plane Block (ESPB) arm to data from electronic health records (EHR) of patients who had not received the ESPB. The EHR data was never obtained, so no comparison was conducted.
Arm/Group | Erector Spinae Plane Block (ESPB) | External control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT05625802/Prot_SAP_000.pdf